CLINICAL TRIAL: NCT05933759
Title: Weight Reduction With the Low-Insulin-Method in an Occupational Health Setting
Brief Title: Weight Reduction With the Low-Insulin-Method
Acronym: WeR-LIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West German Center of Diabetes and Health (Other)
Collaborators: University of Bonn (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: WeR-LIM
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Lifestyle intervention with education via the Low-Insulin-App, low-carb diet, self-monitoring of weight and steps, and telemedical coaching.
  Interventions: Behavioral: Telemedical coaching; Behavioral: Low-Insulin-Method
- Control group (Active Comparator): Lifestyle intervention with education via the Low-Insulin-App, low-carb diet, self-monitoring of weight and steps.
  Interventions: Behavioral: Low-Insulin-Method

INTERVENTIONS:
Behavioral: Telemedical coaching — Individual telemedical coaching delivered by a nutritional consultant
  Arms: Intervention group
Behavioral: Low-Insulin-Method — Lifestyle intervention with education via the Low-Insulin-App, low-carb diet, self-monitoring of weight and steps

SUMMARY:
Background: Overweight and obesity affect health, quality of life and ability to work. Therefore, the Low-Insulin-Method was developed to support overweight and obese people in weight loss.

Method: In a randomized controlled clinical trial, the effect of the lifestyle intervention program 'Low-Insulin-Method', delivered by the Low-Insulin-App including low-carb diet, self monitoring of weight, physical activity and telemedical coaching is examined compared to a control group without coaching. The learning contents are taught in 30 videos and 5 online meetings. The intervention group additionally gets 4 individual care calls. The state of health is examined at the beginning and after 12 weeks.

Objective: The aim is to develop a training and counseling program for overweight or obese individuals with diabetes risk or type 2 diabetes, which can be used both for primary and for tertiary prevention of overweight-related diseases.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index 25 kg/m2

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Weight change in kg | 12 weeks
  Estimated treatment difference

SECONDARY OUTCOMES:
body mass index in kg/m2 | 12 weeks
  Estimated treatment difference
waist circumference in cm | 12 weeks
  Estimated treatment difference
hip circumference in cm | 12 weeks
  Estimated treatment difference
fat mass in kg | 12 weeks
  Estimated treatment difference
lean body mass in kg | 12 weeks
  Estimated treatment difference
muscle mass in kg | 12 weeks
  Estimated treatment difference
energy expenditure in kcal | 12 weeks
  Estimated treatment difference
blood pressure in mmHg | 12 weeks
  Estimated treatment difference
quality of life (short form questionnaire) in units on a scale | 12 weeks
  Estimated treatment difference minimum 0, maximum 100 higher scores mean a better outcome
depression (German version of the Center for Epidemiological Studies-Depression Scale) in units on a scale | 12 weeks
  Estimated treatment difference minimum 0, maximum 100 higher scores mean a worse outcome
physical activity in min/day | 12 weeks
  Estimated treatment difference
physical activity in steps/day | 12 weeks
  Estimated treatment difference
eating behaviour (German version of the Three-factor Eating Questionnaire) in units on a scale | 12 weeks
  Estimated treatment difference minimum 0, maximum 100 higher scores mean a better outcome
total cholesterol in mg/dl | 12 weeks
  Estimated treatment difference
HDL cholesterol in mg/dl | 12 weeks
  Estimated treatment difference
LDL cholesterol in mg/dl | 12 weeks
  Estimated treatment difference
triglycerides in mg/dl | 12 weeks
  Estimated treatment difference
fasting blood glucose in mg/dl | 12 weeks
  Estimated treatment difference
insulin in µU/ml | 12 weeks
  Estimated treatment difference
HbA1c in % | 12 weeks
  Estimated treatment difference
food frequency (German version of the food frequency questionnaire) in units on a scale | 12 weeks
  Estimated treatment difference minimum 0, maximum 100 higher scores mean a better outcome

OTHER OUTCOMES:
gut microbiome composition in percent | 12 weeks
  difference between groups

CONTACTS AND LOCATIONS:
Locations (1):
- West German Centre of Diabetes and Health, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No